CLINICAL TRIAL: NCT05086250
Title: A Prospective, Single Center, Double Blind, Randomized, Crossover Feasibility Study of Oral Ketamine Versus Placebo for the Treatment of Anxiety in Patients With Pancreatic Cancer
Brief Title: Feasibility Study of Oral Ketamine Versus Placebo for the Treatment of Anxiety in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Scott A. Irwin, MD, PhD, Director, Patient and Family Support Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIT2019-18-IRWIN-KETANX
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Pancreatic Cancer
Keywords: ketamine; placebo
MeSH Terms: conditions — Anxiety Disorders; Pancreatic Neoplasms | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, research staff, or subjects. The following study procedures will be in place to ensure double-blind administration of study treatments.
  * Access to the randomization code will be strictly controlled
  * Packaging and labeling of test and control treatments will be identical to maintain the blind The research pharmacist will manage the investigational agent. The blind will be maintained through the effort of the research pharmacist and the pharmacy. Unblinding will only occur when it is deemed medically necessary. The date and reason for breaking the blind will be documented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Ketamine Followed by Placebo (Experimental): Weekly oral administration of 0.5mg/kg ketamine for 4 weeks, followed by weekly oral administration of placebo for 4 weeks (separated by a washout period of 2 weeks).
  Interventions: Drug: Ketamine; Drug: Placebo
- Arm B: Placebo Followed by Ketamine (Experimental): Weekly oral administration of placebo for 4 weeks, followed by weekly oral administration of 0.5mg/kg ketamine for 4 weeks (separated by a washout period of 2 weeks).
  Interventions: Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Weekly oral administration of 0.5mg/kg ketamine for 4 weeks, followed by weekly oral administration of placebo for 4 weeks (separated by a washout period of 2 weeks).
  Other Names: Ketalar
  Arms: Arm A: Ketamine Followed by Placebo
Drug: Placebo — Weekly oral administration of 0.5mg/kg ketamine for 4 weeks, followed by weekly oral administration of placebo for 4 weeks (separated by a washout period of 2 weeks).
  Arms: Arm A: Ketamine Followed by Placebo
Drug: Placebo — Weekly oral administration of placebo for 4 weeks, followed by weekly oral administration of 0.5mg/kg ketamine for 4 weeks (separated by a washout period of 2 weeks).
  Arms: Arm B: Placebo Followed by Ketamine
Drug: Ketamine — Weekly oral administration of placebo for 4 weeks, followed by weekly oral administration of 0.5mg/kg ketamine for 4 weeks (separated by a washout period of 2 weeks).
  Other Names: Ketalar
  Arms: Arm B: Placebo Followed by Ketamine

SUMMARY:
This is a prospective, single center, double blind, randomized, crossover feasibility study of oral ketamine versus placebo for the treatment of anxiety in patients with pancreatic cancer currently receiving or within 12 weeks of receiving cancer targeted therapy. The primary objective is to determine the feasibility of enrolling subjects and treatment adherence. The secondary objectives are to describe the safety and tolerability. Exploratory objectives are to assess the effect of ketamine/placebo on Depression, Anxiety, Physical Function, Pain Interference, Pain Intensity, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities as measured by PROMIS Anxiety Short Form 7a and the PROMIS-29 Profile v2.1 of Patient Reported Outcomes, as well as changes in circulatory inflammatory cytokines, blood glutamine levels, and other biomarkers of anxiety and/or depression.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. Participant has been diagnosed with pancreatic cancer.
3. Receiving or within twelve weeks of having received cancer targeted treatment, including surgery, radiation, chemotherapy, immunotherapy, or other cancer targeted therapy.
4. Age ≥ 18 years.
5. Has moderate to severe anxiety according to the PROMIS Anxiety Short Form 7a and/or PROMIS-29 anxiety module (T-score of > 60).
6. Documented adequate liver function within the screening period.
7. Use of concomitant standard antidepressants targeting anxiety (e.g. SSRIs) is permitted if dose has been the same for at least 12 weeks prior to study entry and patient still meets inclusion #5.
8. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and while receiving study drug. Women of child-bearing potential must have a negative urine or blood pregnancy test at screening. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and study staff immediately.
9. Must be able to read and understand English.
10. Required not to engage in potentially hazardous activities, such as driving a motor vehicle or operating machinery, after receiving a medication dose until the next day after a restful sleep (as per recommendations with Spravato).
11. Agrees to abstain from alcohol use while taking study medication.

Exclusion Criteria:

1. Initial cancer diagnosis ≤6 weeks prior to Day 0.
2. Meets MINI International Neuropsychiatric Interview (MINI Plus), criteria for diagnoses of schizophrenia, bipolar illness, delirium or psychosis.
3. Scores ≥ 10 on the Suicidal Risk Assessment (SRA).
4. History of allergic reactions or hypersensitivity to ketamine.
5. Documented history of severe cardiac insufficiency (NYHA III or IV), with currently uncontrolled and/or unstable cardiac or coronary artery disease.
6. Current or recent significant tachyarrhythmia, severe angina, or myocardial ischemia, as assessed by a study physician.
7. Documented history of poorly controlled hypertension (Systolic Blood Pressure > 180 mmHG or Diastolic Blood Pressure > 100 mmHG twice within a one-month period in last two months), with or without antihypertensives.
8. Women who are pregnant or nursing or expect to become pregnant or start nursing during the expected trial duration, and women of childbearing potential who refuse to use contraceptives to prevent childbearing.
9. Uncontrolled hypo- or hyperthyroidism, as assessed by a study physician.
10. Diagnosis of dementia.
11. Treatment with monoamine oxidase inhibitor (MAOI) within 14 days of Day 0.
12. Aneurysmal vascular disease (including thoracic and abdominal aorta, intracranial and peripheral arterial vessels) or arteriovenous malformation.
13. History of intracerebral hemorrhage.
14. Refusal/inability to comply with inclusion criterion #10 (driving restrictions) and inclusion criterion #11 (alcohol abstinence) during study treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrolling subjects which will be measured by the proportion of patients dropping out of study for any reason prior to the end of treatment visit. | 2 months
  The following will be collected as part of this feasibility measurement:
  * Reasons for dropout.
  * Proportion of patients pre-screened that were potentially eligible for study participation.
  * Proportion of patients that were potentially eligible who were approached.
  * Proportion of approached patients that decline study participation and why.
  * Proportion of approached patients that agreed to participate.
  * Proportion of approached that were randomized.
  * Proportion of patients completing study through End of Treatment visit and each follow-up visit.

SECONDARY OUTCOMES:
To investigate the safety of oral ketamine in patients with pancreatic cancer and anxiety, which will be assessed by the number of adverse events related to study treatment per CTCAE v.5. | 3 months
  Th number of adverse events related to study treatment assessed per CTCAE v.5.
To investigate the tolerability of oral ketamine in patients with pancreatic cancer and anxiety, which will be measured by patient-reported Ketamine Adverse Symptom Checklist and Impact scores. | 3 months
  This is a self-report tool that provides patient rating (none, mild, moderate, severe) of 33 potential side effects of ketamine. The Adverse Symptom Checklist (ASC) is scored 0 (none), mild (1), moderate (2), and severe (3 points). This scale also asks patients to quantify side effect interference in daily activities, also scored the same way (Min value 0, Max Value 3). Therefore, the total score for the ASC has Min value 0, Max 102 where total higher scores mean a worse outcome. The ASC responses will be dichotomized (frequency: 0%-25% vs >25%; intensity: none, mild vs moderate, or greater; burden: none to mild impairment vs moderate or greater impairment) and will be descriptively summarized by each treatment arm at each assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Irwin, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States